CLINICAL TRIAL: NCT06034054
Title: The Effect of Nurse Counselling on Quality of Life, Functional Capacity and Knowledge, Attitudes and Beliefs in Patients With Acute Coronary Syndrome
Brief Title: Acute Coronary Syndrome and Nurse Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iskenderun State Hospital (Other)
Responsible Party: Principal Investigator, Deniz Gülistan ER, Angiography nurse, Iskenderun State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DGulistan-01
Record Dates: First submitted 2023-08-26; First posted 2023-09-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease
Keywords: Acute Coronary Syndrome; Counseling; Nursing
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing counseling (Experimental): The individuals included in nursing counseling group were given counseling by the research nurse for 6 months.
  Interventions: Other: nursing counceling
- Control (No Intervention): Individuals included in control group were followed up routinely in the outpatient clinic for 6 months.

INTERVENTIONS:
Other: nursing counceling — * Providing an educational booklet containing information about pastry, verbally explaining the content of the prepared educational booklet.
  * Answering the information and questions that the patient needs in addition, and receiving contact information in October.
  * Monthly calls will be made to patients 6. providing information that the same tests will be performed again per month, if necessary, this monthly call counseling by reaching out without waiting indicating what they can receive.
  Arms: Nursing counseling

SUMMARY:
The goal of this clinical trial is to examine in patients with acute coronary syndrome. The main questions it aims to answer are:

* Does nurse counseling affect quality of life?
* Does nurse counseling affect functional capacity?
* Does nurse counseling affect knowledge, attitudes and beliefs about syndromes?

Participants will be trained using the training booklet, and nursing counseling will then be provided for six months.

If there is a comparison group: Researchers will compare with the control group to see if the nurse counseling has had an effect.

DETAILED DESCRIPTION:
After obtaining verbal and written consent from the participants, they are required to answer the questions on the Diagnosis Form, Acute Coronary Syndrome Response Index, and Multiple Quality of Life Scale. Then, preliminary measurements will be made and a 6-minute corridor walking test will be applied. While the control group will be followed up routinely, the training booklet prepared for the intervention group will be explained orally. Participants will then be informed that they will be called monthly. They will be told that they can reach these monthly calls and consult the nurse when they need it. After this stage, interviews with patients will begin. The standard way of communication with the participants by the researchers is by telephone, and a total of 6 interviews will be provided, the first of which is in the 1st month after the application of the tests. In each call, all the information in the training booklet will be repeated, additional information will be given in line with the needs and demands of the person, their questions will be answered and the interview will be ended. Although it varies according to the individual interviewed, it is predicted that these telephone interviews will last for 30 minutes on average. Apart from these standard calls, individuals in need will be able to reach the researcher face-to-face during phone calls, text messages, instant messaging methods or hospital visits, and in this way, the counseling process will continue actively for 6 months. After six months, the final tests will be done.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old, diagnosed with Acute Coronary Syndrome and treated with a stent,
* Treatment preventing communication is not a problem, literate,
* There is no obstacle to performing the 6-minute walk test.
* who did not accept to participate, were included in the study.

Exclusion Criteria:

* <18 years of age,
* Mental or cognitive impairment,
* Diagnosed with SpO2 <80,
* Peripheral arterial disease, lower extremity amputation, impaired tumor or open wound of lower extremity, and deep vein thrombosis, 6 munites corridor Walk test Parts of individuals who are contraindicated in making are not included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Life quality | 6 mounth
  Multidimensional index of life quality will be applied(This scale is the "multidimensional quality of life scale", the Turkish validity and reliability of which was established in 2012.)
Functional capacity | 6 mounth
  Functional Capacity Evaluation Form will be applied.
Acute Coronary Syndromes | 6 mount
  Acute Coronary Syndrome Response Index will be applied.It was translated into Turkish and a reliability and validity study was conducted in 2016. A questionnaire consisting of 33 items was applied to evaluate the knowledge, attitudes and beliefs of individuals with acute coronary syndrome regarding the disease.

CONTACTS AND LOCATIONS:
Overall Officials: sevgin samancıoğlu bağlama, assoc.prof, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- İskenderun State Hospital, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No